CLINICAL TRIAL: NCT06331234
Title: Determination of the Effects of Vena Cava Inferior Measurements on Acute Kidney Injury and Mortality During Intensive Care Admission.
Brief Title: Effects of Vena Cava Inferior Measurements on AKI and Mortality.
Status: Not yet recruiting | Type: Observational
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Ayse Belin Ozer, Prof. Dr., Inonu University
Other Study IDs: VCI
Record Dates: First submitted 2024-03-20; First posted 2024-03-26 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Intensive Care Unit; Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Vena cava inferior diameter — he VExUS score is obtained as follows: VEXUS 0: IVC < 20mm; VEXUS 1: IVC ≥ 20mm with normal patterns or mild abnormalities; VEXUS 2: IVC ≥ 20mm with severe abnormality in at least one pattern and VEXUS 3: IVC ≥ 20mm and severe abnormalities in multiple patterns.
  Other Names: VEXUS score

SUMMARY:
Fluid overload is harmful in critically ill patients; In addition to increasing mortality, it may increase the incidence of acute kidney injury (AKI), length of ICU stay, and duration of mechanical ventilation by causing end-organ damage. (1-3) Mortality attributable to AKI is 20% and is an independent determinant of mortality. (4) Venous load ultrasonography score (VExUS) is a new systemic congestion scoring method based on inferior vena cava dilation and pulsed wave Doppler (PW-Doppler) morphology of the hepatic, portal and renal veins. It has been proposed as a score to assess systemic congestion. When the IVC diameter is < 2 cm, it means there is no congestion and VEXUS is 0. Mild congestion: In addition to the IVC measuring approximately 2 cm, normal patterns such as the systolic wave being greater than the diastolic wave in the hepatic vein PW-doppler, pulsatility below 30% in the portal vein Doppler, continuous flow in the renal vein PW-doppler, or slightly abnormal patterns, i.e. hepatic The systolic wave in vein PW-doppler is smaller than the diastolic wave, the pulsatility in portal PW-doppler is between 30-50%, and the renal vein PW-doppler is accompanied by biphasic flow, and VEXUS is scored as 1. Moderate congestion is scored as VEXUS 2, which is measured as IVC 2 cm or more, plus inversion of the systolic wave on hepatic vein PW-doppler, pulsatility greater than 50% on portal PW-doppler, and discontinuous monophasic flow with only the diastolic phase on renal vein PW-doppler. It is accompanied by one of the serious abnormal patterns such as There is severe congestion, that is, VEXUS 3: IVC diameter of 2 cm or more and the presence of at least two seriously abnormal PW-Doppler morphologies. (5) The primary aim of this study is to describe the prevalence of venous congestion based on VExUS in general ICU patients. Secondary outcomes were to evaluate the association between VExUS, AKI, and 28-day mortality.

DETAILED DESCRIPTION:
In the first 24 hours of hospitalization, the inferior vena cava will be evaluated by an experienced clinician (INTENSIVE CARE SPECIALIST). If the IVC diameter is below 2 cm, the collapsibility index will be checked if the patient is not receiving mechanical ventilation (MV) treatment, and the distensibility index will be checked if the patient is receiving MV treatment. If the IVC diameter is over 2 cm, VEXUS will be performed. As primary outcomes, the development of acute kidney injury within one week and 28-day mortality will be recorded. Acute kidney injury will be performed according to KDIGO criteria. Patients' age, gender, body mass index, comorbidities, medications used before admission to intensive care (especially ACE inhibitors and ARBs), reason for admission to intensive care, fluid therapy applied in the first 24 hours, and fluid balance in the first 24 hours will be recorded. In patients taken from the emergency department, the amount of fluid taken and removed in the emergency room will also be recorded. Additionally, the use of vasopressors/vasodilators, inotropes, diuretics, colloids and blood products will be recorded. The central venous pressure of patients with a central venous catheter will also be recorded on the first day.

Patients will undergo transthoracic echocardiography and lung ultrasonography simultaneously, and ejection fraction and TAPSE will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a life expectancy of more than 24 hours >18 age

Exclusion Criteria:

* Poor abdominal echogenicity age < 18 postoperative patients, intoxications, life expectancy is less than 24 hours, pregnancy, intraperitoneal pressure > 15 mm Hg, obstructive renal failure or suspected, presence of renal artery stenosis, patients who have had liver and kidney transplants, Presence of liver and kidney tumors, patients receiving dialysis treatment, single kidney and other kidney abnormalities, presence of acute mesenteric ischemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to intensive care
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
acute kidney injury | 7 days
mortality | 28 days
  in 28 days mortality

IPD SHARING:
Plan to Share IPD: Undecided